CLINICAL TRIAL: NCT04329988
Title: Primary Care Validation in French of a Single-question Screening Test for Unhealthy Alcohol Use.
Acronym: DECORA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0889
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2021-01

CONDITIONS: Unhealthy Alcohol Use
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary care patients aged 18 or more: All patients consulting in a general practitioner office, aged 18 or more, who completed the questionnaire
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — A questionnaire will be made available to all eligible patients in general practitioners waiting rooms. This questionnaire will be composed by the single question, followed by the AUDIT and FACE questionnaires, and three socio-demographic questions. This questionnaire will be anonymous. Patients who agree to fill out a questionnaire will place it in a sealed box once completed.

SUMMARY:
Unhealthy alcohol use (UAU) is a very important public health concern. In France UAU is the second cause of avoidable death after tobacco smoking. In 2014, 31% of the French adult population presented with unhealthy alcohol use. Primary care practitioners have access to validated questionnaires in French such as the Alcohol Use Disorder Identification Test (AUDIT) and the Fast Alcohol Consumption Evaluation (FACE). These tests are not often used because of their length.

In 2009 a study by Smith et al in the USA compared a single question with the AUDIT-c (a short version of the AUDIT). The single question was "How many times in the past year have you had X or more drinks in a day?" Where X is 7 for men and 6 for women. This study found that the single question had a comparable sensitivity and a specificity, respectively 81,8% and 79,3%.

The aim of the study is to validate this question in French. First the question has been translated from English to French following the WHO method. The aim of the present study is to validate the French translation by comparing it with the AUDIT and the FACE. A questionnaire will be given to patients with inclusion criteria in general practitioners waiting rooms (15 different locations). This questionnaire will be composed of the single question, followed by the AUDIT and FACE, and three socio-demographic questions. The questionnaire will be anonymous.

ELIGIBILITY:
Inclusion Criteria:

* Consulting in a general practitioner's office
* Over 18 years Old

Exclusion Criteria:

* Less than 18 years old
* Pregnant women or breast-feeding mothers
* People under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population consulting in a primary care office over 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
sensitivity of the single question | At inclusion (Patients will answer the questionnaire only once while waiting in theirs doctor's waiting room).
  sensitivity of the single question as measured versus the AUDIT (Alcohol use disorder identification test) Sensitivity = TP/(TP+FN) TP : true positives : people answering 1 or more at the single question and having a score of 8 or more with the AUDIT questionnaire FN : False Negatives : people answering 0 at the single question and having a score of 8 or more with the AUDIT questionnaire TN : True negatives : people answering 0 at the single question and having a score of 7 or less with the AUDIT questionnaire
specificity of the single question | At inclusion (Patients will answer the questionnaire only once while waiting in theirs doctor's waiting room).
  specificity of the single question as measured versus the AUDIT (Alcohol use disorder identification test).
  Specificity = TN/(TN+FP) TP : true positives : people answering 1 or more at the single question and having a score of 8 or more with the AUDIT questionnaire TN : True negatives : people answering 0 at the single question and having a score of 7 or less with the AUDIT questionnaire FP : False positives : people answering 1 or more at the single question and having a score of 7 or less with the AUDIT questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Cabinet de Médecine Générale Dr Christine Maynie-François, Saint-Quentin-Fallavier, France

IPD SHARING:
Plan to Share IPD: No